CLINICAL TRIAL: NCT00905554
Title: Warm Water Irrigation Versus Standard Air Insufflation for Unsedated Colonoscopy: a Randomized Controlled Trial
Brief Title: Warm Water for Unsedated Colonoscopy
Acronym: WW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Vittorio Terruzzi, MD, Valduce Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WW01
Record Dates: First submitted 2009-05-15; First posted 2009-05-20 (Estimated); Results first posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-09

CONDITIONS: Colonoscopy
Keywords: sedation; warm water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- warm water (Experimental): warm water irrigation during the insertion phase of colonoscopy
  Interventions: Procedure: warm water irrigation
- air (Active Comparator): air insufflation during the insertion phase of colonoscopy
  Interventions: Procedure: air insufflation

INTERVENTIONS:
Procedure: warm water irrigation — warm water irrigation during insertion phase of colonoscopy
  Arms: warm water
Procedure: air insufflation — air insufflation during the insertion phase of colonoscopy
  Arms: air

SUMMARY:
Unsedated colonoscopy is characterized by lower costs, recovery time and incidence of drug-related side effects, although it may be painful for the patient. Based on recent reports, the investigators designed this randomized controlled trial hypothesizing that the use of water irrigation versus air insufflation during the insertion phase of colonoscopy might increase the global tolerability of the examination and the proportion of patients undergoing complete colonoscopy without sedation.

ELIGIBILITY:
Inclusion Criteria:

* adult outpatients willing to undergo colonoscopy without routine initial sedation

Exclusion Criteria:

* refuse to initiate colonoscopy without routine sedation
* inadequate bowel preparation
* incapacity to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Valduce Hospital, Como, CO, Italy

REFERENCES:
- [Derived] Radaelli F, Paggi S, Amato A, Terruzzi V. Warm water infusion versus air insufflation for unsedated colonoscopy: a randomized, controlled trial. Gastrointest Endosc. 2010 Oct;72(4):701-9. doi: 10.1016/j.gie.2010.06.025. PMID 20883846

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical clinic since march 2009 until sample size was reached
Pre-assignment Details: no patient excluded from the study flow after being allocated in the study or control arm
Period: Overall Study
Arm/Group | Warm Water | Air Insufflation
Started | 116 | 114
Completed | 116 | 114
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Warm Water | Air Insufflation | Total
Number analyzed (Participants) | 116 | 114 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 108 | 109 | 217
  >=65 years | 6 | 4 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 58.4 (11.5) | 58.8 (13.3) | 58.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 48 | 96
  Male | 68 | 66 | 134
Region of Enrollment [Number; unit: participants]
  Italy | 116 | 114 | 230

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Undergoing Complete Unsedated Colonoscopy
Time Frame: 6-9 months
Measure: Number; unit: participants
Arm/Group | Warm Water | Air Insufflation
Number analyzed (Participants) | 116 | 114
participants | 101 | 89

2. Secondary Outcome: Evaluation of Pain and Tolerability Scores
Description: Entity of pain and tolerability level on a visual analogic scale (ranging from 0 - no pain, optimal tolerability - to 100 mm - worst pain ever, unbearable)
Time Frame: 6-9 months
Measure: Median (Inter-Quartile Range); unit: Scores on a VAS scale
Arm/Group | Warm Water | Air Insufflation
Number analyzed (Participants) | 116 | 114
Scores on a VAS scale | 28 [12 to 44] | 39 [14 to 54]

ADVERSE EVENTS:
Arm/Group | Warm Water | Air Insufflation
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/114
Other Adverse Events (participants affected / at risk) | 0/116 | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No